CLINICAL TRIAL: NCT02488018
Title: Investigation of Ethiopian Honey: Botanical Origin, Physicochemical, Antioxidant, Microbial Quality, Glycemic Index and Sensory Properties
Brief Title: Investigation of the Glycemic Index of Ethiopian Honey
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Abera Belay, PhD Candidate, Addis Ababa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Honey-1
Record Dates: First submitted 2015-06-27; First posted 2015-07-02 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-07

CONDITIONS: Hyperglycemia, Postprandial
Keywords: Glycemic index; honey; reference glucose
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Provision of experimental honeys (Experimental): Eight experimental monofloral honeys and reference glucose
  Interventions: Biological: Provision of experimental honey

INTERVENTIONS:
Biological: Provision of experimental honey — Acacia, Becium grandiflorum, Croton macrostachys, Eucalyptus globules, Hypoestes, Leaucas abyssinica, Schefflera abyssinica, Syzygium guineense and reference glucose were used as test food.
  25g available carbohydrate of the test food was provided to ten human subjects after fasted for 11 hours overnight.
  Other Names: Honey Glycemic Index

SUMMARY:
The purpose of this study is to determine which of the Ethiopian honeys slowly/rapidly raise the blood glucose level.

DETAILED DESCRIPTION:
Addis Ababa University, College of Natural Sciences, Research Institutional Review Board (IRB) approved this study. Written consent forms were obtained from all 14 volunteers (7 females and 7 males). The subjects were randomly recruited from twenty eight 3rd year Food Science and Postharvest Technology students. People volunteering to participate in the study were excluded if they are: overweight, dieting, smoking, a family history of diabetes, pregnant, metabolic disorders, suffering from any illness or food allergy and regularly taking medication. The participants were checked for glucose tolerance according to the WHO (World Health Organization) classification (fasting glucose <7 mmol/L(millimole per lite) and 2-hour blood glucose concentration after a 25g glucose load <7.8 mmol/L). Ten (5 females and 5 males) were selected from fourteen using lottery sampling methods. Reference glucose and monofloral honeys were used as experimental foods. To determine the GI value, 25 grams of available carbohydrate was fed for ten healthy people in the morning after they have fasted for 11 hours overnight. After fasting blood sample was obtained. The study participants were consumed each honey and reference glucose served. Additional blood samples were taken at 15, 30, 45, 60, 90 and 120 minutes after eating commenced. Blood glucose response (Area under the curve, AUCt) for test food was compared to the blood glucose response of reference glucose (AUCr). AUC was calculated using SAS (Statistical Analysis Software), 2002. Glycemic index (GI) was calculated using:

GI= AUCt/AUCr*100

Where:

AUCt = Area Under the Curve for honey; AUCr = Area Under the Curve for the reference glucose

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes Disease
* Must be able to drink the honeys and reference glucose

Exclusion Criteria:

* Overweight, dieting, smoking, a family history of diabetes, pregnant, metabolic disorders, suffering from any illness or food allergy and regularly taking medication.

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abera Belay, PhDCandidate, Principal Investigator — Addis Ababa University; Gulelat Haki, Professor, Study Chair — Department of Food Science and Technology, Botswana College of Agriculture, University of Botswana.; Kaleab Baye, Asst Prof., Study Chair — Addis Ababa University; Samuel Melaku, Assoc Prof., Study Chair — Columbus State University

IPD SHARING:
Plan to Share IPD: Undecided
Due to the Ethical issue, sharing data to 3rd party is not decided yet.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After a through orientation on research objectives to 3rd year Food Science & Technology students, 14 volunteer free of: overweight, dieting, smoking, family history of diabetes, pregnant, metabolic disorders, and suffering from food allergy were selected. Out of 14 eligible students, 5female and 5male students were selected using lottery sampling.
Pre-assignment Details: The Addis Ababa University, College of Natural Sciences, Research Institutional Review Board (IRB) approved this study. Written consent forms were obtained from all 14 volunteers (7 females and 7 males).
Groups:
- Honey Glycemic Index: Study participants were given 25g available carbohydrate of reference glucose or monofloral honeys of Acacia, Becium grandiflorum, Croton macrostachys, Eucalyptus globules, Hypoestes, Leaucas abyssinica, Schefflera abyssinica, Syzygium guineense in 250 mL of water, after they have fasted for 11 hours overnight.
  Monofloral honeys, namely: collected from honey productive areas; and reference glucose were used as a test food. 25g available carbohydrate of the test foods was provided to all ten human subjects after fasted for 11 hours overnight. After fasting blood sample was collected from the finger. Additional blood samples were taken at 15, 30, 45, 60, 90 and 120 minutes. Glucose concentration of blood samples was used to draw a two-hour blood glucose response curve. Area under curve (AUC) for test food and reference glucose was calculated by trapezoidal rule.
Period: Overall Study
Arm/Group | Honey Glycemic Index
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Provision of Experimental Honeys: Monofloral honeys, namely: Acacia, Becium grandiflorum, Croton macrostachys, Eucalyptus globules, Hypoestes, Leaucas abyssinica, Schefflera abyssinica, Syzygium guineense collected from honey productive areas; and reference glucose were used as a test food. 25g available carbohydrate of the test foods was provided to all ten human subjects after fasted for 11 hours overnight. After fasting blood sample was collected from the finger. Additional blood samples were taken at 15, 30, 45, 60, 90 and 120 minutes. Glucose concentration of blood samples was used to draw a two-hour blood glucose response curve. Area under curve (AUC) for test food and reference glucose was calculated by trapezoidal rule.
Arm/Group | Provision of Experimental Honeys
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.60 (1.17)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Blood glucose level (mmol/L) [Number; unit: Participant] — Participants with a blood glucose level of <7 mmol/L after fasting (0 time)
  Participant | 10

OUTCOME MEASURES:

1. Primary Outcome: Examine Effect of Monofloral Honey Types on Glycemic Index of Health Human Subjects
Description: Ten healthy individuals consumed monofloral honeys (25g of available carbohydrate in 250 mL water) after fasting for 11 hours. Blood glucose levels (mmol/L) were recorded at 0, 15, 30, 45, 60, 90 and 120 minutes. Time (0, 15, 30, 45, 60, 90 and 120 minutes) verse blood glucose levels (mmol/L) used to establish the area under the curve (AUC) for the honeys and reference glucose. This was used to calculate the glycemic index of honey each honey (GI= AUC for honey/AUC for reference glucose*100). All 10 participants took eight different honeys and reference glucose on nine different days (with randomized allocation of samples).
Time Frame: 36 days (9 tests in 4 days interval)
Population: All 10 participants took, 25g available carbohydrate of eight different honeys and reference glucose, on nine different days in 4 days interval. Blood was taken from finger prick using automatic lancet at 0, 15, 30, 45, 60, 90 and 120 minutes; glucose levels were recorded and area under the blood glucose curve was calculated.
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Provision of Experimental Honeys: Monofloral honeys, namely: Acacia, Becium grandiflorum, Croton macrostachys, Eucalyptus globules, Hypoestes, Leaucas abyssinica, Schefflera abyssinica, Syzygium guineense collected from honey productive areas; and reference glucose were used as a test food.
  25g available carbohydrate of the test foods was provided to ten human subjects after fasted for 11 hours overnight. After fasting blood sample was collected from the finger. Additional blood samples were taken at 15, 30, 45, 60, 90 and 120 minutes. Glucose concentration of blood samples was used to draw a two-hour blood glucose response curve. Area under curve (AUC) for test food and reference glucose was calculated by trapezoidal rule.
Arm/Group | Provision of Experimental Honeys
Number analyzed (Participants) | 10
Index
  Acacia | 54.73 (7.19)
  Becium grandiflorum | 62.82 (7.73)
  Croton macrostachyus | 60.31 (7.26)
  Eucalyptus globulus | 59.54 (7.34)
  Hypoestes | 63.22 (6.69)
  Leucas abyssinica | 64.06 (7.58)
  Schefflera abyssinica | 71.90 (7.47)
  Syzygium guineense | 63.07 (7.37)
Statistical Analysis 1: Comparison: Provision of Experimental Honeys; Hypothesis Ho: Honey plant origin does not affects the glycemic index of human subjects. Ha: Honey plant origin affects the glycemic index of human subjects; Test type: Superiority or Other; p < 0.01, ANOVA; Degree of freedom for the model (treatment) was 8

ADVERSE EVENTS:
Time Frame: Total Number of participants Affected: 0 Total Number of participants at Risk: 10
Groups:
- Honey Glycemic Index: Study participants were given 25g available carbohydrate of reference glucose or honey in 250 mL of water, after they have fasted for 11 hours overnight.
Arm/Group | Honey Glycemic Index
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No